CLINICAL TRIAL: NCT00617708
Title: A Phase I and Randomized Phase II Trial of Gemcitabine + Erlotinib (NSC-718781) + IMC-A12 (NSC-742460) vs. Gemcitabine + Erlotinib as First-Line Treatment in Patients With Metastatic Pancreatic Cancer
Brief Title: S0727 Gemcitabine Hydrochloride and Erlotinib Hydrochloride With or Without Monoclonal Antibody Therapy in Treating Patients With Metastatic Pancreatic Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00797; NCI-2009-00797 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000586427; SWOG-S0727; S0727 (Other: Southwest Oncology Group); S0727 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 2008-02-15; First posted 2008-02-18 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — cixutumumab; Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (erlotinib, gemcitabine, cixutumumab) (Experimental): Patients receive erlotinib hydrochloride PO once daily on days 1-28, gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15, and cixutumumab IV over 60 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cixutumumab; Drug: erlotinib hydrochloride; Drug: gemcitabine hydrochloride
- Arm II (erlotinib, gemcitabine) (Active Comparator): Patients receive erlotinib hydrochloride and gemcitabine hydrochloride as in arm I. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Biological: cixutumumab — Given IV
  Other Names: anti-IGF-1R recombinant monoclonal antibody IMC-A12; IMC-A12
  Arms: Arm I (erlotinib, gemcitabine, cixutumumab)
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar

SUMMARY:
This randomized phase I/II trial is studying the side effects and best dose of monoclonal antibody therapy when given together with gemcitabine hydrochloride and erlotinib hydrochloride and to see how well they work compared with giving gemcitabine hydrochloride and erlotinib hydrochloride alone as first-line therapy in treating patients with metastatic pancreatic cancer that cannot be removed by surgery. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving erlotinib hydrochloride and gemcitabine hydrochloride together with monoclonal antibody therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the appropriate dose of IMC-A12 (cixutumumab) to use in combination with gemcitabine (gemcitabine hydrochloride) and erlotinib (erlotinib hydrochloride). (Phase I) II. To assess progression-free survival in patients with metastatic pancreatic cancer treated with IMC-A12 plus gemcitabine and erlotinib compared to those treated with gemcitabine plus erlotinib alone. (Phase II) III. To assess overall survival in each of the two treatment arms in this group of patients. (Phase II) IV. To assess the total response probability (confirmed and unconfirmed, complete and partial responses) in each of the two treatment arms in the subset of this group of patients with measurable disease. (Phase II) V. To assess the qualitative and quantitative toxicities in each of the two treatment arms in this group of patients. (Phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study of cixutumumab followed by a randomized, phase II study.

Patients are initially enrolled into the phase I portion of the study to determine the recommended phase II dose (RPTD) of cixutumumab. Once the RPTD is determined, patients are enrolled into the phase II portion of the study.

PHASE I (LIMITED INSTITUTIONS): Patients receive erlotinib hydrochloride orally (PO) once daily on days 1-28, gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1, 8, and 15, and cixutumumab IV over 60 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

PHASE II (ALL SWOG MEMBERS): Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive erlotinib hydrochloride, gemcitabine hydrochloride, and cixutumumab at the RPTD as in phase I.

ARM II: Patients receive erlotinib hydrochloride and gemcitabine hydrochloride as in arm I.

In both arms, treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Previously collected tumor tissue is obtained for gene expression analyses by RT-PCR, RNA isolation, and cDNA synthesis. Blood samples are collected periodically for correlative studies. Samples are assessed for the potential relationship between gene expression levels, germline polymorphisms, Ras and P13K mutations and progression-free survival and overall survival.

After completion of study treatment, patients are followed every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed pancreatic adenocarcinoma

  * Stage IV disease (any T, any N, M1 [distant metastases])
  * Unresectable disease
  * Histologic diagnosis based on a metastatic site must be compatible with pancreatic cancer
* Measurable and/or nonmeasurable disease
* No endocrine or neuroendocrine tumors, lymphoma of the pancreas, or ampullary cancer
* No macroscopic residual disease post-resection as the only site of disease
* No clinically significant ascites
* No known brain metastases

  * Patients with neurologic signs or symptoms must undergo brain imaging studies AND studies must be negative for disease
* Zubrod performance status 0-1
* ANC ≥ 1,500/mcL
* Platelet count ≥ 100,000/mcL
* Hemoglobin ≥ 9 g/dL
* Leukocytes ≥ 3,000/mcL
* Total bilirubin normal
* SGOT or SGPT ≤ 2.5 times upper limit of normal (ULN)
* Serum creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Fasting serum glucose < 120 mg/dL or below the ULN

  * Patients with diabetes mellitus who meet this criterion must be on a stable dietary or therapeutic regimen for this condition
* INR ≤ 1.5 and PTT ≤ 5 seconds above ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Willing to submit previously collected tumor tissue specimens
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to anti-IGF-1R recombinant monoclonal antibody IMC-A12
* No active acute or chronic infections requiring antibiotics
* No significant ongoing cardiac problems, including any of the following:

  * Myocardial infarction within the past 6 months
  * Uncontrolled hypertension
  * Unstable angina
  * Uncontrolled arrhythmia
  * Congestive heart failure
* No known HIV infection
* No other prior malignancy, except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Adequately treated stage I or II cancer from which the patient is currently in complete remission
  * Any other cancer from which the patient has been disease-free for 5 years
* At least 14 days since prior surgery
* At least 28 days since prior radiotherapy for palliation to metastatic sites

  * Patient must have other untreated metastatic sites that would qualify them for this protocol
* At least 6 months since prior adjuvant chemotherapy
* No prior chemotherapy, hormonal therapy, immunotherapy, or chemoradiotherapy for advanced or locally advanced pancreatic cancer, including drugs that target either EGFR or IGFR
* No plans to receive concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or any other type of therapy for treatment of cancer
* No prior gemcitabine hydrochloride
* No prior chimerized or murine monoclonal antibody therapy
* No concurrent CYP3A4 inducers including, but not limited to, any of the following:

  * Rifampicin
  * Rifabutin
  * Rifapentine
  * Phenytoin
  * Carbamazepine
  * Phenobarbital
  * Hypericum perforatum (St. John's wort)
* No concurrent CYP3A4 inhibitors including, but not limited to, any of the following:

  * Atazanavir
  * Clarithromycin
  * Indinavir
  * Itraconazole
  * Ketoconazole
  * Nefazodone
  * Nelfinavir
  * Ritonavir
  * Saquinavir
  * Telithromycin
  * Troleandomycin
  * Voriconazole
* Concurrent prophylactic low-dose coumadin or low molecular weight heparin allowed provided coagulation criteria are met
* Full-dose anticoagulation allowed provided coagulation criteria are met and are under strict control and monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2008-03; Primary Completion 2012-09-01 (Actual); Study Completion 2014-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Philip, Principal Investigator — SWOG Cancer Research Network
Locations (146):
- United States (146):
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - City of Hope Medical Center, Duarte, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Marin General Hospital, Greenbrae, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - University of Southern California, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons Inc, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - University of California Medical Center At Irvine-Orange Campus, Orange, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - California Pacific Medical Center, San Francisco, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Well Star Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Joseph's-Candler Health System, Savannah, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Wayne State University, Detroit, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Mercy Health Partners-Mercy Campus, Muskegon, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Liberty Radiation Oncology Clinic, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Arnot Ogden Medical Center, Elmira, New York
  - Highland Hospital, Rochester, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Veterans Administration Medical Center - Cincinnati, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Saint Luke's Episcopal Hospital, Houston, Texas
  - Veterans Administration Medical Center, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Memorial Hospital Of Martinsville, Martinsville, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison Bremerton Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology and Oncology PLLC, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Oncology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health Cooperative, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Ph I: Erlotinib + Gemcitabine + IMC-A12; Ph II: Erlotinib + Gemcitabine + IMC-A12: Erlotinib 100 mg PO once daily, Gemcitabine 1,000 mg/m^2 IV days 1, 8 and 15, and IMC-A12 6 mg/kg IV days 1, 8, 15 and 22. One cycle = 28 days.
- Ph II: Erlotinib + Gemcitabine: Erlotinib 100 mg PO once daily, Gemcitabine 1,000 mg/m^2 IV days 1, 8 and 15. One cycle = 28 days.
Period: Overall Study
Arm/Group | Ph I: Erlotinib + Gemcitabine + IMC-A12 | Ph II: Erlotinib + Gemcitabine + IMC-A12 | Ph II: Erlotinib + Gemcitabine
Started | 10 | 60 | 64
Eligible and Began Protocol Therapy | 9 | 57 | 59
Completed | 0 | 0 | 0
Not Completed | 10 | 60 | 64
Not completed — Adverse Event | 0 | 6 | 9
Not completed — Withdrawal by Subject | 1 | 1 | 7
Not completed — Death | 0 | 6 | 5
Not completed — Progression/Relapse | 7 | 40 | 36
Not completed — Not protocol specified | 1 | 4 | 2
Not completed — Not eligible | 1 | 3 | 5

BASELINE CHARACTERISTICS:
Population: Eligible patients who began protocol therapy
Groups:
- Total: Total of all reporting groups
Arm/Group | Ph I: Erlotinib + Gemcitabine + IMC-A12 | Ph II: Erlotinib + Gemcitabine + IMC-A12 | Ph II: Erlotinib + Gemcitabine | Total
Number analyzed (Participants) | 9 | 57 | 59 | 125
Age, Continuous [Median (Full Range); unit: years] | 61 [39 to 82] | 63 [36 to 87] | 64 [42 to 82] | 63 [35 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 34 | 25 | 62
  Male | 6 | 23 | 34 | 63
Race/Ethnicity, Customized [Number; unit: participants]
  White | 5 | 44 | 51 | 100
  Black | 2 | 10 | 6 | 18
  Asian | 1 | 2 | 2 | 5
  Unknown | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 1 | 3 | 5 | 9
  Non-Hispanic | 8 | 53 | 47 | 108
  Unknown | 0 | 1 | 7 | 8

OUTCOME MEASURES:

1. Secondary Outcome: Overall Survival
Description: From date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Up to 3 years
Population: Eligible patients in the Phase II portion of the study.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Erlotinib + Gemcitabine + IMC-A12: Erlotinib 100 mg PO once daily, Gemcitabine 1,000 mg/m^2 IV days 1, 8 and 15, and IMC-A12 6 mg/kg IV days 1, 8, 15 and 22. One cycle = 28 days.
- Erlotinib + Gemcitabine: Erlotinib 100 mg PO once daily, Gemcitabine 1,000 mg/m^2 IV days 1, 8 and 15. One cycle = 28 days.
Arm/Group | Erlotinib + Gemcitabine + IMC-A12 | Erlotinib + Gemcitabine
Number analyzed (Participants) | 57 | 59
months | 7.0 [4.2 to 8.9] | 6.5 [5.0 to 7.7]

2. Primary Outcome: Maximum Tolerated Dose Determination
Description: Maximum dose of IMC-A12 (in combination with erlotinib and gemcitabine) at which 3/10 or fewer patients have dose-limiting toxicities (DLT). Toxicities graded according to the NCI Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE 3.0). DLT apply only during cycle 1 and should be drug-related (possible, probable, or definite).
Time Frame: 28 days
Population: Phase I patients receiving at least three doses of the assigned dose during Cycle 1 or whom developed a DLT.
Measure: Number; unit: mg/kg IMC-A12
Arm/Group | Ph I: Erlotinib + Gemcitabine + IMC-A12
Number analyzed (Participants) | 10
mg/kg IMC-A12 | 6

3. Secondary Outcome: Response
Description: Confirmed response (CR) is two or more objective statuses of CR a minimum of four weeks apart documented before progression or symptomatic deterioration. Partial response (PR) is two or more objective statuses of PR or better a minimum of four weeks apart documented before progression or symptomatic deterioration. Unconfirmed CR is one objective status of CR documented before progression or symptomatic deterioration but not qualifying as CR or PR. Unconfirmed PR is one objective status of PR documented before progression or symptomatic deterioration but not qualifying as CR, PR or unconfirmed CR.
Time Frame: Up to 3 years
Population: Eligible patients in the Phase II portion of the study with measurable disease and adequate response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib + Gemcitabine + IMC-A12 | Erlotinib + Gemcitabine
Number analyzed (Participants) | 51 | 53
percentage of participants | 13.7 [5.7 to 26.3] | 15.3 [7.2 to 27.0]

4. Secondary Outcome: Toxicity
Description: Number of patients with Grade 3 through 5 adverse events that are related to study drug. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 3 years
Population: Eligible patients who received any treatment and were assessed for toxicity were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Ph I: Erlotinib + Gemcitabine + IMC-A12 | Ph II: Erlotinib + Gemcitabine + IMC-A12 | Ph II: Erlotinib + Gemcitabine
Number analyzed (Participants) | 9 | 57 | 57
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 0 | 9 | 4
  AST, SGOT | 0 | 6 | 3
  Acidosis (metabolic or respiratory) | 0 | 1 | 0
  Adult respiratory distress syndrome (ARDS) | 0 | 0 | 1
  Albumin, serum-low (hypoalbuminemia) | 0 | 3 | 0
  Alkaline phosphatase | 0 | 4 | 3
  Allergic reaction/hypersensitivity | 1 | 0 | 0
  Anorexia | 1 | 7 | 6
  Bilirubin (hyperbilirubinemia) | 0 | 5 | 0
  Calcium, serum-low (hypocalcemia) | 0 | 1 | 1
  Cardiac troponin I (cTnI) | 0 | 3 | 0
  Cardiac-ischemia/infarction | 0 | 0 | 1
  Cardiopulmonary arrest, cause unknown (non-fatal) | 0 | 0 | 1
  Dehydration | 3 | 6 | 5
  Diarrhea | 2 | 3 | 2
  Dizziness | 0 | 1 | 0
  Dysphagia (difficulty swallowing) | 0 | 0 | 1
  Dyspnea (shortness of breath) | 0 | 2 | 4
  Edema: limb | 0 | 0 | 1
  Edema: trunk/genital | 0 | 0 | 1
  Fatigue (asthenia, lethargy, malaise) | 4 | 16 | 12
  GGT (gamma-glutamyl transpeptidase) | 0 | 1 | 0
  Glucose, serum-high (hyperglycemia) | 2 | 16 | 1
  Hemoglobin | 0 | 9 | 8
  Hypotension | 0 | 3 | 1
  Hypoxia | 0 | 1 | 2
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 0 | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - UTI | 0 | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Bil. tree | 0 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 1 | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 0 | 1 | 2
  Inf w/normal ANC or Gr 1-2 neutrophils - Pancreas | 0 | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Skin | 0 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 0 | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils -Up aerodig | 0 | 1 | 0
  Infection-Other (Specify) | 0 | 1 | 0
  Left ventricular systolic dysfunction | 0 | 1 | 0
  Leukocytes (total WBC) | 1 | 9 | 5
  Liver dysfunction/failure (clinical) | 0 | 0 | 1
  Lymphatics-Other (Specify) | 0 | 0 | 1
  Lymphopenia | 1 | 4 | 5
  Magnesium, serum-low (hypomagnesemia) | 0 | 1 | 0
  Mucositis/stomatitis (functional/symp) - Oral cav | 0 | 1 | 0
  Muscle weakness, not d/t neuropathy - Extrem-lower | 0 | 1 | 0
  Muscle weakness, not d/t neuropathy - body/general | 0 | 5 | 3
  Nausea | 4 | 9 | 6
  Neuropathy: sensory | 0 | 1 | 0
  Neutrophils/granulocytes (ANC/AGC) | 3 | 21 | 10
  Obstruction, GI - Duodenum | 0 | 0 | 1
  Opportunistic inf associated w/gt=Gr 2 lymphopenia | 1 | 0 | 0
  PTT (Partial thromboplastin time) | 0 | 1 | 0
  Pain - Abdomen NOS | 0 | 0 | 1
  Pain - Eye | 0 | 1 | 0
  Pain - Head/headache | 0 | 1 | 0
  Pain - Muscle | 0 | 0 | 1
  Pancreas, exocrine enzyme deficiency | 0 | 1 | 0
  Pancreatic endocrine: glucose intolerance | 0 | 6 | 0
  Pericardial effusion (non-malignant) | 0 | 0 | 1
  Personality/behavioral | 0 | 1 | 0
  Platelets | 2 | 16 | 7
  Pleural effusion (non-malignant) | 0 | 0 | 1
  Pneumonitis/pulmonary infiltrates | 0 | 1 | 2
  Potassium, serum-low (hypokalemia) | 0 | 1 | 1
  Pulmonary/Upper Respiratory-Other (Specify) | 0 | 1 | 1
  Rash/desquamation | 0 | 0 | 1
  Rash: acne/acneiform | 0 | 3 | 2
  Rash: erythema multiforme | 0 | 1 | 0
  SVT and nodal arrhythmia - Atrial fibrillation | 0 | 1 | 0
  Sodium, serum-low (hyponatremia) | 1 | 5 | 1
  Stricture/stenosis (incl anastomotic), Stomach | 0 | 0 | 1
  Syncope (fainting) | 0 | 3 | 0
  Thrombosis/embolism (vascular access-related) | 0 | 1 | 0
  Thrombosis/thrombus/embolism | 0 | 4 | 1
  Tremor | 0 | 1 | 0
  Uric acid, serum-high (hyperuricemia) | 0 | 1 | 0
  Ventricular arrhythmia - Ventricular fibrillation | 0 | 1 | 0
  Vision-blurred vision | 0 | 1 | 0
  Vision-photophobia | 0 | 1 | 0
  Vomiting | 2 | 5 | 1
  Weight loss | 0 | 2 | 0

5. Primary Outcome: Progression-Free Survival
Description: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression free are censored at date of last contact.
Time Frame: Up to 3 years
Population: Eligible patients in the Phase II portion of the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib + Gemcitabine + IMC-A12 | Erlotinib + Gemcitabine
Number analyzed (Participants) | 57 | 59
months | 3.6 [2.4 to 5.3] | 3.6 [1.8 to 5.3]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Ph I: Erlotinib + Gemcitabine + IMC-A12 | Ph II: Erlotinib + Gemcitabine + IMC-A12 | Ph II: Erlotinib + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 5/9 | 34/57 | 33/57
Other Adverse Events (participants affected / at risk) | 9/9 | 56/57 | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ph I: Erlotinib + Gemcitabine + IMC-A12 (N=9) | Ph II: Erlotinib + Gemcitabine + IMC-A12 (N=57) | Ph II: Erlotinib + Gemcitabine (N=57)
Hemoglobin (Blood and lymphatic system disorders) | 0 | 6 | 2
Lymphatics-Other (Specify) (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrioventricular block - first degree (Cardiac disorders) | 0 | 1 | 0
Cardiac-ischemia/infarction (Cardiac disorders) | 0 | 1 | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (non-malignant) (Cardiac disorders) | 0 | 0 | 1
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Ventricular arrhythmia - Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0
Ascites (non-malignant) (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 0 | 0 | 1
Hemorrhage, GI - Duodenum (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 0 | 1 | 1
Ileus, GI (functional obstruction of bowel) (Gastrointestinal disorders) | 0 | 0 | 1
Incontinence, anal (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 3
Obstruction, GI - Duodenum (Gastrointestinal disorders) | 0 | 0 | 1
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 1 | 0 | 1
Obstruction, GI - Stomach (Gastrointestinal disorders) | 0 | 1 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 0 | 9 | 3
Vomiting (Gastrointestinal disorders) | 2 | 4 | 3
Death not associated with CTCAE term - Death NOS (General disorders) | 0 | 1 | 0
Edema: limb (General disorders) | 0 | 1 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 | 3 | 4
Hepatobiliary/Pancreas-Other (Specify) (Hepatobiliary disorders) | 0 | 2 | 0
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 0 | 0 | 1
Portal vein flow (Hepatobiliary disorders) | 0 | 0 | 1
Stricture/stenosis (incl anastomotic)-Biliary tree (Hepatobiliary disorders) | 0 | 0 | 2
Allergic reaction/hypersensitivity (Immune system disorders) | 1 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 0 | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Ab NOS (Infections and infestations) | 1 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Bil. tree (Infections and infestations) | 0 | 1 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 1 | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Catheter (Infections and infestations) | 0 | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 0 | 1 | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Pancreas (Infections and infestations) | 0 | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Perit cav (Infections and infestations) | 0 | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 0 | 2 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 0 | 1 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 0 | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils -Up aerodig (Infections and infestations) | 0 | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils-Foreign bod (Infections and infestations) | 0 | 1 | 0
Infection with unknown ANC - Blood (Infections and infestations) | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 0 | 1 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 | 1 | 1
AST, SGOT (Investigations) | 0 | 1 | 2
Alkaline phosphatase (Investigations) | 0 | 1 | 2
Amylase (Investigations) | 0 | 1 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 0 | 5 | 2
Cardiac troponin I (cTnI) (Investigations) | 0 | 2 | 1
Creatinine (Investigations) | 1 | 1 | 0
Lipase (Investigations) | 0 | 1 | 0
Lymphopenia (Investigations) | 0 | 1 | 0
Pancreas, exocrine enzyme deficiency (Investigations) | 0 | 1 | 0
Platelets (Investigations) | 0 | 2 | 0
Weight loss (Investigations) | 0 | 1 | 0
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 | 1 | 0
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 6 | 5
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 | 4 | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 1 | 2
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 3 | 0
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 0 | 5 | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 9 | 10
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Neuropathy: motor (Nervous system disorders) | 0 | 1 | 0
Syncope (fainting) (Nervous system disorders) | 0 | 2 | 0
Confusion (Psychiatric disorders) | 1 | 2 | 0
Mood alteration - agitation (Psychiatric disorders) | 0 | 1 | 0
Personality/behavioral (Psychiatric disorders) | 0 | 1 | 0
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 0 | 1 | 0
Incontinence, urinary (Renal and urinary disorders) | 0 | 1 | 0
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 2 | 3
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 5 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ph I: Erlotinib + Gemcitabine + IMC-A12 (N=9) | Ph II: Erlotinib + Gemcitabine + IMC-A12 (N=57) | Ph II: Erlotinib + Gemcitabine (N=57)
Hemoglobin (Blood and lymphatic system disorders) | 8 | 38 | 39
Cardiac Arrhythmia-Other (Specify) (Cardiac disorders) | 1 | 0 | 0
Cardiac-ischemia/infarction (Cardiac disorders) | 1 | 0 | 0
SVT and nodal arrhythmia - Atrial tachycardia/PAT (Cardiac disorders) | 1 | 0 | 0
SVT and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Auditory/Ear-Other (Specify) (Ear and labyrinth disorders) | 2 | 0 | 0
Dry eye syndrome (Eye disorders) | 1 | 4 | 0
Ocular/Visual-Other (Specify) (Eye disorders) | 1 | 0 | 0
Vision-blurred vision (Eye disorders) | 0 | 5 | 4
Vision-flashing lights/floaters (Eye disorders) | 3 | 3 | 0
Constipation (Gastrointestinal disorders) | 7 | 33 | 27
Diarrhea (Gastrointestinal disorders) | 5 | 32 | 27
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 0 | 3
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 | 6 | 5
Flatulence (Gastrointestinal disorders) | 0 | 3 | 5
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 0 | 3 | 5
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 | 10 | 4
Hemorrhage, GI - Abdomen NOS (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 4 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 3
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1 | 17 | 0
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 2 | 10 | 4
Nausea (Gastrointestinal disorders) | 9 | 43 | 34
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 1 | 0 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 5 | 17 | 21
Pain - Oral cavity (Gastrointestinal disorders) | 0 | 4 | 0
Pain - Rectum (Gastrointestinal disorders) | 1 | 0 | 0
Pain - Stomach (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 26 | 25
Edema: limb (General disorders) | 1 | 12 | 16
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8 | 47 | 43
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 3 | 5 | 15
Pain - Chest/thorax NOS (General disorders) | 0 | 3 | 0
Pain-Other (Specify) (General disorders) | 0 | 7 | 3
Rigors/chills (General disorders) | 1 | 5 | 7
Allergic reaction/hypersensitivity (Immune system disorders) | 0 | 0 | 3
Allergy/Immunology-Other (Specify) (Immune system disorders) | 0 | 3 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Ab NOS (Infections and infestations) | 1 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 2 | 3 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 1 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 1 | 0 | 0
Infection-Other (Specify) (Infections and infestations) | 0 | 3 | 3
Opportunistic inf associated w/gt=Gr 2 lymphopenia (Infections and infestations) | 1 | 0 | 0
Bruising (in absence of Gr 3-4 thrombocytopenia) (Injury, poisoning and procedural complications) | 2 | 0 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 8 | 34 | 30
AST, SGOT (Investigations) | 8 | 36 | 31
Alkaline phosphatase (Investigations) | 5 | 35 | 25
Bilirubin (hyperbilirubinemia) (Investigations) | 3 | 18 | 18
Creatinine (Investigations) | 3 | 9 | 8
INR (of prothrombin time) (Investigations) | 0 | 4 | 7
Leukocytes (total WBC) (Investigations) | 4 | 29 | 29
Lymphopenia (Investigations) | 1 | 8 | 10
Metabolic/Laboratory-Other (Specify) (Investigations) | 0 | 5 | 4
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 6 | 30 | 20
PTT (Partial thromboplastin time) (Investigations) | 0 | 3 | 4
Platelets (Investigations) | 9 | 42 | 36
Weight loss (Investigations) | 3 | 27 | 25
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 | 25 | 18
Anorexia (Metabolism and nutrition disorders) | 5 | 35 | 31
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 | 0 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 | 18 | 14
Dehydration (Metabolism and nutrition disorders) | 2 | 12 | 11
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 9 | 27 | 29
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 | 7 | 4
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 | 5 | 5
Pancreatic endocrine: glucose intolerance (Metabolism and nutrition disorders) | 0 | 7 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 | 4 | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 | 11 | 4
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 | 10 | 15
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 | 19 | 19
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 2 | 10 | 9
Pain - Back (Musculoskeletal and connective tissue disorders) | 2 | 13 | 8
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Pain - Joint (Musculoskeletal and connective tissue disorders) | 3 | 7 | 3
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6 | 7
Dizziness (Nervous system disorders) | 2 | 8 | 7
Neuropathy: sensory (Nervous system disorders) | 1 | 9 | 4
Ocular/Visual-Other (Specify) (Nervous system disorders) | 1 | 0 | 0
Pain - Head/headache (Nervous system disorders) | 1 | 6 | 0
Syncope (fainting) (Nervous system disorders) | 0 | 3 | 0
Taste alteration (dysgeusia) (Nervous system disorders) | 3 | 21 | 16
Tremor (Nervous system disorders) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 3 | 0
Insomnia (Psychiatric disorders) | 2 | 10 | 12
Mood alteration - agitation (Psychiatric disorders) | 1 | 0 | 0
Mood alteration - anxiety (Psychiatric disorders) | 1 | 11 | 8
Mood alteration - depression (Psychiatric disorders) | 3 | 8 | 5
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 0 | 0 | 3
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 5 | 0
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 | 0 | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 12 | 8
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 | 15 | 20
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 0
Mucositis/stomatitis (clinical exam) - Pharynx (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 0 | 5 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 13 | 10
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 | 4 | 10
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 8 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 | 12 | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 | 14 | 22
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 6 | 31 | 24
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 | 6 | 6
Hypertension (Vascular disorders) | 1 | 4 | 4
Hypotension (Vascular disorders) | 3 | 6 | 5
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less